CLINICAL TRIAL: NCT04950179
Title: Peritoneal Dialysis-Related Infection Rates and Outcomes of Antibiotic Treatments Among Continuous Ambulatory Peritoneal Dialysis Patients at a Tertiary University Hospital: A 5-Year Retrospective Study
Brief Title: PDRI Rates Among CAPD Patients at a Tertiary University Hospital: A 5-Year Retrospective Study
Status: Completed | Type: Observational
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Collaborators: Silpakorn University (Other)
Responsible Party: Sponsor
Other Study IDs: PDRI-2020
Record Dates: First submitted 2021-06-25; First posted 2021-07-06 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Peritoneal Dialysis-related Infection
Keywords: Peritoneal dialysis-related infection; Infectious peritonitis; Exit-site infection; Tunnel infection; Infection rate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PDRI patients — The study was conducted by retrospective data collection from medical records of 135 continuous ambulatory peritoneal dialysis (CAPD) patients at Phramongkutklao Hospital from January 1, 2016 to December 31, 2020.

SUMMARY:
Peritoneal dialysis-related infection is a complication that leads to peritoneal dialysis catheter removal or patient death. The present study aimed to investigate peritoneal dialysis-related infection rates, causative pathogens, appropriation of antibiotic use, treatment outcomes and trend in antimicrobial resistance of causative pathogens.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were at least 18 years old.
2. Patients who were diagnosed with stage 5 chronic kidney disease (eGFR < 15 ml/min/1.73m^2).
3. Patients who were undergoing Continuous Ambulatory Peritoneal Dialysis (CAPD) at CAPD clinic, Phramongkutklao Hospital during January 1, 2016 to December 31, 2020.

Exclusion Criteria:

1. Patients with incomplete data records that invalid to include in the process of data analysis
2. Patients who were not treated and started their first CAPD at CAPD clinic, Phramongkutklao Hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were undergoing Continuous Ambulatory Peritoneal Dialysis (CAPD) at CAPD clinic, Phramongkutklao Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Rate of peritoneal dialysis-related infection | January 1, 2016 to December 31, 2020
  Retrospective data collection from patients' medical records
Treatment outcomes of peritoneal dialysis-related infection | January 1, 2016 to December 31, 2020
  Retrospective data collection from patients' medical records

SECONDARY OUTCOMES:
Causative pathogens of peritoneal dialysis-related infection | January 1, 2016 to December 31, 2020
  Retrospective data collection from patients' medical records
Appropriation of antibiotic use in the treatments of peritoneal dialysis-related infection | January 1, 2016 to December 31, 2020
  Retrospective data collection from patients' medical records

CONTACTS AND LOCATIONS:
Overall Officials: Pamila Tasanavipas, MD, Study Chair — Phramongkutklao Hospital and College of Medicine; Daraporn Rungprai, BCP, Study Director — Faculty of Pharmacy, Silpakorn University; Vorada Pengsong, Principal Investigator — Faculty of Pharmacy, Silpakorn University; Vattanai Dhamnimitchok, Principal Investigator — Faculty of Pharmacy, Silpakorn University; Vilai Wisuthip, Principal Investigator — Faculty of Pharmacy, Silpakorn University; Supichaya Hluangbumroong, Principal Investigator — Faculty of Pharmacy, Silpakorn University
Locations (1):
- Phramongkutklao Hospital, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luvira V, Satirapoj B, Supasyndh O, Chaiprasert A, Ruangkanchanasetr P, Nata N, Kanjanakul I, Supaporn T, Choovichian P, Bijaphala S, Luvira U, Phiboonbanakit D. A single-centre experience: peritoneal dialysis-related infections in patients on long-term dialysis. J Med Assoc Thai. 2011 Sep;94 Suppl 4:S30-6. PMID 22043564
- [Background] Kanjanabuch T, Chancharoenthana W, Katavetin P, Sritippayawan S, Praditpornsilpa K, Ariyapitipan S, Eiam-Ong S, Dhanakijcharoen P, Lumlertgul D. The incidence of peritoneal dialysis-related infection in Thailand: a nationwide survey. J Med Assoc Thai. 2011 Sep;94 Suppl 4:S7-12. PMID 22043560
- [Background] Perl J, Fuller DS, Bieber BA, Boudville N, Kanjanabuch T, Ito Y, Nessim SJ, Piraino BM, Pisoni RL, Robinson BM, Schaubel DE, Schreiber MJ, Teitelbaum I, Woodrow G, Zhao J, Johnson DW. Peritoneal Dialysis-Related Infection Rates and Outcomes: Results From the Peritoneal Dialysis Outcomes and Practice Patterns Study (PDOPPS). Am J Kidney Dis. 2020 Jul;76(1):42-53. doi: 10.1053/j.ajkd.2019.09.016. Epub 2020 Jan 10. PMID 31932094
- [Background] Wang HH, Huang CH, Kuo MC, Lin SY, Hsu CH, Lee CY, Chiu YW, Chen YH, Lu PL. Microbiology of peritoneal dialysis-related infection and factors of refractory peritoneal dialysis related peritonitis: A ten-year single-center study in Taiwan. J Microbiol Immunol Infect. 2019 Oct;52(5):752-759. doi: 10.1016/j.jmii.2018.10.013. Epub 2019 Jan 8. PMID 30665844
- [Background] Chen HC, Shieh CC, Sung JM. Increasing Staphylococcus Species Resistance in Peritoneal Dialysis-Related Peritonitis over a 10-Year Period in a Single Taiwanese Center. Perit Dial Int. 2018 Jul-Aug;38(4):266-270. doi: 10.3747/pdi.2017.00226. PMID 29987065
- [Background] Li PK, Szeto CC, Piraino B, Bernardini J, Figueiredo AE, Gupta A, Johnson DW, Kuijper EJ, Lye WC, Salzer W, Schaefer F, Struijk DG; International Society for Peritoneal Dialysis. Peritoneal dialysis-related infections recommendations: 2010 update. Perit Dial Int. 2010 Jul-Aug;30(4):393-423. doi: 10.3747/pdi.2010.00049. No abstract available. PMID 20628102
- [Background] Szeto CC, Li PK, Johnson DW, Bernardini J, Dong J, Figueiredo AE, Ito Y, Kazancioglu R, Moraes T, Van Esch S, Brown EA. ISPD Catheter-Related Infection Recommendations: 2017 Update. Perit Dial Int. 2017 Mar-Apr;37(2):141-154. doi: 10.3747/pdi.2016.00120. No abstract available. PMID 28360365
- [Background] Li PK, Szeto CC, Piraino B, de Arteaga J, Fan S, Figueiredo AE, Fish DN, Goffin E, Kim YL, Salzer W, Struijk DG, Teitelbaum I, Johnson DW. ISPD Peritonitis Recommendations: 2016 Update on Prevention and Treatment. Perit Dial Int. 2016 Sep 10;36(5):481-508. doi: 10.3747/pdi.2016.00078. Epub 2016 Jun 9. No abstract available. PMID 27282851